CLINICAL TRIAL: NCT05646706
Title: Effect and Safety of Semaglutide 7.2 mg Once-weekly in Participants With Obesity
Brief Title: A Research Study to See How Semaglutide Helps People With Excess Weight, Lose Weight (STEP UP)
Acronym: STEP UP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4999; U1111-1274-4259 (Other: World Health Organization (WHO)); 2022-000790-94 (EudraCT Number)
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Semaglutide 7.2 mg (Experimental): Participants will receive once-weekly injection of semaglutide subcutaneously (s.c.) in 20 week dose escalation period with dose escalation (0.25 milligram [mg], 0.5 mg, 1.0 mg, 1.7 mg, 2.4 mg, and 7.2 mg) every fourth week. Treatment was continued on the maintenance dose of 7.2 mg once-weekly for an additional 52 weeks until week 72.
  Interventions: Drug: Semaglutide
- Semaglutide 2.4 mg (Experimental): Participants will receive once-weekly s.c. injection of semaglutide in 20 week dose escalation period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, and 2.4 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. Treatment was continued on the maintenance dose of 2.4 mg once-weekly for an additional 52 weeks until week 72.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive once-weekly s.c. injection of placebo matched to semaglutide for 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Participants will receive once-weekly s.c. injections of semaglutide in escalating doses (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, 2.4 mg and 7.2 mg) every fourth week. Treatment was continued on the maintenance dose of 7.2 mg once-weekly for an additional 52 weeks. Injections may be administered in the thigh, abdomen, or upper arm, at any time of day irrespective of meals.
  Arms: Semaglutide 7.2 mg
Drug: Semaglutide — Participants will receive once-weekly s.c. injections of semaglutide in escalating doses (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, and 2.4 mg) every fourth week. Treatment was continued on the maintenance dose of 2.4 mg once-weekly for an additional 52 weeks. Injections may be administered in the thigh, abdomen, or upper arm, at any time of day irrespective of meals.
  Arms: Semaglutide 2.4 mg
Drug: Placebo — Participants will receive once-weekly s.c. injection of placebo matched to semaglutide for 72 weeks. Injections may be administered in the thigh, abdomen, or upper arm, at any time of day irrespective of meals.
  Arms: Placebo

SUMMARY:
This study will look at how much weight participants will lose from the start to the end of the study. The weight loss in participants taking the investigational high dose of semaglutide will be compared to the weight loss in people taking "dummy" medicine and a lower dose of semaglutide. In addition to taking the medicine, participants will have talks with study staff about healthy food choices and how to be more physically active. Participants will either get semaglutide or "dummy" medicine. Which treatment participants get is decided by chance. Participants are more likely (4 out of 5) to get semaglutide than the "dummy" medicine. The study medicine will be injected briefly, under skin, with a thin needle, typically in the stomach, thighs, or upper arms. In the first part of the study, participants will get one injection once a week until they reach the planned dose. The second part of the study, which might last a couple of months, is a transition period, where participant will get three injections, taken right after each other, once a week. The duration of the study intervention (trial product and lifestyle intervention) will be 72 weeks followed by a 9-week follow-up period without study interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age above or equal to 18 years at the time of signing informed consent.
* Body mass index (BMI) greater than or equal to 30.0 kilogram per square meter (kg/m^2).
* History of at least one self-reported unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

* HbA1c greater than or equal to 48 millimoles per mole (mmol/mol) (6.5 percent) as measured by the central laboratory at screening.
* History of type 1 or type 2 diabetes.
* Treatment with glucose-lowering agent(s) within 90 days before screening.
* A self-reported change in body weight greater than 5 kilograms (kg) (11 pounds) within 90 days before screening irrespective of medical records.
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1407 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Semaglutide 7.2 mg versus Placebo: Relative change in body weight | From baseline (week 0) to end of treatment (week 72)
  Measured in percentage (%).
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction greater than or equal to (>=) 5% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.

SECONDARY OUTCOMES:
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction >=10% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction >=15% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction >=20% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction >=25% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Change in waist circumference | From baseline (week 0) to end of treatment (week 72)
  Measured in centimeters (cm).
Semaglutide 7.2 mg versus Semaglutide 2.4 mg: Relative change in body weight | From baseline (week 0) to end of treatment (week 72)
  Measured in percentage (%).
Semaglutide 7.2 mg versus Semaglutide 2.4 mg: Number of participants who achieve body weight reduction >=20% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Semaglutide 2.4 mg: Number of participants who achieve body weight reduction >=25% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Change in body weight | From baseline (week 0) to end of treatment (week 72)
  Measured in kilograms (kg).
Semaglutide 7.2 mg versus Placebo: Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 72)
  Measured in kilogram per square meter (kg/m^2).
Semaglutide 7.2 mg versus Placebo: Change in total fat mass (%) | From baseline (week 0) to end of treatment (week 72)
  Measured in percentage (%).
Semaglutide 7.2 mg versus Placebo: Change in total fat mass (liters) | From baseline (week 0) to end of treatment (week 72)
  Measured in liters.
Semaglutide 7.2 mg versus Placebo: Change in lean body mass (%) | From baseline (week 0) to end of treatment (week 72)
  Measured in percentage (%).
Semaglutide 7.2 mg versus Placebo: Change in lean body mass (liters) | From baseline (week 0) to end of treatment (week 72)
  Measured in liters.
Semaglutide 7.2 mg versus Placebo: Change in visceral fat mass (%) | From baseline (week 0) to end of treatment (week 72)
  Measured in percentage (%).
Semaglutide 7.2 mg versus Placebo: Change in visceral fat mass (liters) | From baseline (week 0) to end of treatment (week 72)
  Measured in liters.
Semaglutide 7.2 mg versus Placebo: Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 72)
  Measured in millimeters of mercury (mmHg).
Semaglutide 7.2 mg versus Placebo: Change in diastolic blood pressure | From baseline (week 0) to end of treatment (week 72)
  Measured in mmHg.
Semaglutide 7.2 mg versus Placebo: Change in total cholesterol | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in triglycerides | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in free fatty acids | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in high-sensitivity c reactive protein (hsCRP) | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Number of participants with change in lipid-lowering treatment (decrease, no change, increase) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of participants with change in antihypertensive treatment (decrease, no change, increase) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 72)
  Measured in percentage (%).
Semaglutide 7.2 mg versus Placebo: Change in fasting plasma glucose | From baseline (week 0) to end of treatment (week 72)
  Measured in milligrams per deciliter (mg/dL).
Semaglutide 7.2 mg versus Placebo: Change in fasting serum insulin | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Number of participants with change in glycaemic category (Normo-glycaemia, pre-diabetes, type 2 diabetes [T2D]) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of adverse events (AEs) | From baseline (week 0) to end of study (week 81)
  Measured as count of events.
Semaglutide 7.2 mg versus Placebo: Number of serious adverse events (SAEs) | From baseline (week 0) to end of study (week 81)
  Measured as count of events.
Semaglutide 7.2 mg versus Placebo: Change in pulse | From baseline (week 0) to end of treatment (week 72)
  Measured in beats per minute (bmp).
Semaglutide 7.2 mg versus Semaglutide 2.4 mg: Number of AEs | From baseline (week 0) to end of study (week 81)
  Measured as count of events.
Semaglutide 7.2 mg versus Semaglutide 2.4 mg: Number of SAEs | From baseline (week 0) to end of study (week 81)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (106):
- United States (21):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Chambliss Clinical Trials, LLC, Montgomery, Alabama
  - Healthscan Clinical Trials,LLC., Montgomery, Alabama
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - Florida Inst For Clin Res LLC, Orlando, Florida
  - Florida Institute For Clinical Research LLC, Orlando, Florida
  - East West Med Res Inst, Honolulu, Hawaii
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - AMC Community Endocrinology, Albany, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Elligo Clin Res Centre, Austin, Texas
  - Velocity Clin Res, Dallas, Dallas, Texas
  - UT Southwestern Medical Center-CRU, Dallas, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Sugar Lakes Family Practice PA, Sugar Land, Texas
  - National Clin Res Inc., Richmond, Virginia
  - Selma Medical Associates, Winchester, Virginia
- Bulgaria (10):
  - Medical centre Zdrave 1 OOD, Kozloduy
  - Medical center Hippocrates Lukovit EOOD, Lukovit
  - IPMC - Dr. Elizabeta Dimitrova, Petrich
  - Medical center Smolyan clinical research OOD, Smolyan
  - DCC Ascendent OOD, Sofia
  - SGHAT Dr. Shterev EOOD, Sofia
  - Acibadem City Clinic MHAT Tokuda Department of Endocrinology and Metabolic Diseases, Sofia
  - Medical Centre Medical Arts Medico-dental centre, Sofia
  - Medical Center Medical Plus EOOD, Varna
  - AIPSMC Dr. Evelina Zlatanova EOOD, Varna
- Canada (7):
  - Ocean West Research Clinic, Surrey, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Hamilton Med Res Group, Hamilton, Ontario
  - Milestone Research, London, Ontario
- Czechia (7):
  - Ordinace praktického lékaře, Benátky Na Jizerou
  - Edumed Broumov, Broumov
  - Fakultní nemocnice Královské Vinohrady_Praha 10, Prague
  - Endocare, Prague
  - Institut klinické a experimentalni mediciny, Prague
  - Poliklinika Michnova - Obezitologie, Prague
  - Fledip s.r.o., Prague
- Germany (10):
  - Medizinisches Versorgungszentrum Am Bahnhof Spandau GbR, Berlin
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - Praxis Dr. med. M. Esser, Essen
  - Zentrum für klinische Forschung, Dr. med. Lüdemann, Falkensee
  - MedicalCenter am Clemenshospital - Schwerpunktpraxis für Diabetologie und Ernährungsmedizin, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Praxis Dr. med. Wenzl-Bauer, Rehlingen-Siersburg
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
  - Forschungszentrum Ruhr KliFoCenter GmbH, Kahrmann, Witten
- Greece (9):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - Gen Hospital of Athens Laiko,1st Dpt. of Propaedeutic Inter, Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - General Hospital of Lamia, Lamia
  - General Hospital of Thessaloniki 'G. Gennimatas, Thessaloniki
  - AHEPA General University Hospital, Thessaloniki
  - "Ippokrateio" G.H. of Thessaloniki, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
- Hungary (7):
  - Lausmed Kft., Baja, Bács-Kiskun county
  - Belinus Bt., Debrecen, Hajdú-Bihar
  - Borbánya Praxis E.Ü. Kft., Nyíregyháza, Szabolcs-Szatmar Varmegye
  - ClinDiab Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Bajcsy-Zsilinszky Kórház, Budapest
  - MED-TIMA Kft., Budapest
  - Fejér Megyei Szent György Oktatókórház, Székesfehérvár
- Norway (3):
  - Falck Norge AS, Hamar
  - Oslo universitetssykehus HF Aker, Oslo
  - Sykehuset i Vestfold HF, Tønsberg, Tønsberg
- Poland (8):
  - Med. Cent. Diabet. Endo. Metabol. DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - NZOZ Przychodnia Specjalistyczna Medica, Lublin, Lubelski
  - NZOZ "CenterMed Lublin" Sp. z o.o., Lublin, Lublin Voivodeship
  - Kresmed Sp. z o. o., Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne SUM w Katowicach, Katowice
  - NBR Polska Tomasz Klodawski, Warsaw
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw
- Portugal (6):
  - Unidade Local De Saude De Matosinhos E.P.E., Senhora Da Hora, Matosinhos, Matosinhos
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Unidade Local De Saude De Lisboa Ocidental E.P.E. - Hospital Egas Moniz, Lisbon
  - Hospital Da Luz S.A., Lisbon
  - Unidade Local de Saude de Sao Joao E.P.E, Porto
  - Hospital Luz Arrabida, S.A., Vila Nova de Gaia
- Slovakia (8):
  - MUDr. Dagmar Prokesova, Endokrinologicka ambulancia, Bratislava
  - MEDIMAD, s.r.o., Endokrinologicka ambulancia, Bratislava
  - IN-DIA s.r.o., Lučenec
  - SIN AZUCAR s.r.o., Malacky
  - MED-CENTRUM, s.r.o., Martin
  - SVAJDLEROVA, s.r.o., Prešov
  - MEDIVASA, s.r.o., Angiologicka ambulancia, Žilina
  - Dom srdca, s.r.o., Žilina
- South Africa (10):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Medi-Clinic Bloemfontein, Bloemfontein, Free State
  - Soweto Clinical Trial Centre, Johannesburg, Gauteng
  - Deepak Lakha, Johannesburg, Gauteng
  - Hemant Makan, Johannesburg, Gauteng
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Precise Clinical Solutions (Pty) Ltd, Durban, KwaZulu-Natal
  - Dr N.K. Gounden Medical Centre, Durban, KwaZulu-Natal
  - Lenmed Shifa Private Hospital, Durban, KwaZulu-Natal
  - Dr T Padayachee, eMkhomazi, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisktrials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Wharton S, Freitas P, Hjelmesaeth J, Kabisch M, Kandler K, Lingvay I, Quiroga M, Rosenstock J, Garvey WT; STEP UP trial group. Once-weekly semaglutide 7.2 mg in adults with obesity (STEP UP): a randomised, controlled, phase 3b trial. Lancet Diabetes Endocrinol. 2025 Nov;13(11):949-963. doi: 10.1016/S2213-8587(25)00226-8. Epub 2025 Sep 14. PMID 40961952